CLINICAL TRIAL: NCT01989117
Title: Prospective Non-randomized Comparative Study Evaluating the Effectiveness of Osteopathy in the Preoperative Treatment of Postoperative Pain in Patients Undergoing Total Knee Replacement in Osteoarthritis Indication
Brief Title: Effectiveness of Osteopathy in the Preoperative Treatment of Postoperative Pain in Patients Undergoing Total Knee Replacement
Status: Completed | Type: Observational
Sponsor: Hospital Ambroise Paré Paris (Other)
Responsible Party: Principal Investigator, Shahnaz Klouche, MD, Physician Responsible of Clinical Research, Hospital Ambroise Paré Paris
Other Study IDs: APR102013
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Total Knee Replacement; Osteoarthritis of the Knee; Preoperative Osteopathic Care
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Osteopathy
- No osteopathy

SUMMARY:
Osteopathy is an alternative healthcare that seems effective in relieving the pain of patients. The main purpose of this study is to evaluate the efficacy of preoperative osteopathic care in patients undergoing total knee arthroplasty (TKA) for osteoarthritis. The secondary objectives are to assess pain during the first postoperative month on a VAS and knee function and quality of life at 6 months and 1 year. Our hypothesis is that osteopathy will decrease postoperative pain and increase knee function.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee arthroplasty (TKA)
* For osteoarthritis of the knee
* Without surgical history on the operated knee

Exclusion Criteria:

* Previous surgery on the operated knee
* Bilateral TKA
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for primary total knee arthroplasty (TKA) for osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Self-assessment of knee pain on Visual Analog Scale (VAS) | At one month postoperatively

SECONDARY OUTCOMES:
Pain self-assessment during the first postoperative month on Visual analog scale (VAS) | Twice daily during the first postoperative month
Functional assessment of the knee with International Knee Society (IKS) score | At six months postoperatively
Functional assessment of the knee with International Knee Society (IKS) score | At one year postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Ambroise Pare, Boulogne-Billancourt, France